CLINICAL TRIAL: NCT02142738
Title: A Randomized Open-Label Phase III Trial of Pembrolizumab Versus Platinum Based Chemotherapy in 1L Subjects With PD-L1 Strong Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Pembrolizumab (MK-3475) Compared to Platinum-Based Chemotherapies in Participants With Metastatic Non-Small Cell Lung Cancer (MK-3475-024/KEYNOTE-024)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-024; 142728 (Registry Identifier: JAPIC); MK-3475-024 (Other: Merck Protocol Number); 2014-000323-25 (EudraCT Number)
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-05

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: Programmed cell death-1 (PD-1); Programmed cell death 1 (PD1); Programmed death-ligand 1 (PDL1); PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Paclitaxel; Carboplatin; Pemetrexed; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg, administered as intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Drug: Pembrolizumab
- Paclitaxel+Carboplatin (Active Comparator): Participants receive paclitaxel 200 mg/m^2 and carboplatin Area Under the Curve (AUC) 5 or 6, administered as IV infusion on Day 1 of each 21-day cycle for 4-6 cycles followed by optional pemetrexed 500 mg/m^2 every three weeks (Q3W) maintenance for participants with non-squamous histologies for the remainder of the study or until documented PD or participant discontinuation. If PD occurs, participants may be able to receive pembrolizumab Q3W in a second course of treatment.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Pemetrexed
- Pemetrexed+Carboplatin (Active Comparator): Participants receive pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6, IV infusion on Day 1 of each 21-day cycle for 4-6 cycles; participants with non-squamous histologies may then receive pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle as maintenance therapy for the remainder of the study or until documented PD or participant discontinuation. If PD occurs, participants may be able to receive pembrolizumab Q3W in a second course of treatment.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed
- Pemetrexed+Cisplatin (Active Comparator): Participants receive pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, administered as IV infusion on Day 1 of each 21-day cycle for 4-6 cycles followed by optional pemetrexed 500 mg/m^2 Q3W maintenance for the remainder of the study or until documented PD or participant discontinuation. If PD occurs, participants may be able to receive pembrolizumab Q3W in a second course of treatment.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin
- Gemcitabine+Carboplatin (Active Comparator): Participants receive gemcitabine 1250 mg/m^2, administered as IV infusion on Days 1 and 8 of each 21-day cycle and carboplatin AUC 5 or 6, administered as IV infusion on Day 1 of a 21-day cycle, for 4-6 cycles or until documented PD or participant discontinuation. If PD occurs, participants may be able to receive pembrolizumab Q3W in a second course of treatment.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine
- Gemcitabine+Cisplatin (Active Comparator): Participants receive gemcitabine 1250 mg/m^2, administered as IV infusion on Days 1 and 8 of each 21-day cycle and cisplatin 75 mg/m^2, administered as IV infusion on Day 1 of each 21-day cycle for 4-6 cycles or until documented PD or participant discontinuation. If PD occurs, participants may be able to receive pembrolizumab Q3W in a second course of treatment.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab IV solution
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: Paclitaxel — Paclitaxel IV solution
  Arms: Paclitaxel+Carboplatin
Drug: Carboplatin — Carboplatin IV solution
  Arms: Gemcitabine+Carboplatin; Paclitaxel+Carboplatin; Pemetrexed+Carboplatin
Drug: Pemetrexed — Pemetrexed Lyophilized Powder for Infusion
  Arms: Paclitaxel+Carboplatin; Pemetrexed+Carboplatin; Pemetrexed+Cisplatin
Drug: Cisplatin — Cisplatin IV solution
  Arms: Gemcitabine+Cisplatin; Pemetrexed+Cisplatin
Drug: Gemcitabine — Gemcitabine Lyophilized Powder for Infusion
  Arms: Gemcitabine+Carboplatin; Gemcitabine+Cisplatin

SUMMARY:
This is a study to assess the efficacy and safety of pembrolizumab (MK-3475/SCH 900475) compared to standard of care (SOC) platinum-based chemotherapies in the treatment of participants with previously untreated stage IV, programmed cell death ligand 1 (PD-L1) strong expressing Non-Small Cell Lung Cancer (NSCLC). The primary hypothesis of this study is that participants with PD-L1 strong NSCLC will have a longer Progression Free Survival (PFS), as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) when treated with pembrolizumab than when treated with SOC platinum-based chemotherapies.

With Amendment 09 (20 December 2017), once participants have achieved the study objective or the study has ended, participants will be discontinued from this study and enrolled in an extension study to continue protocol-defined assessments and treatment.

DETAILED DESCRIPTION:
Treatment Phase: Participants randomized to pembrolizumab will be treated for up to 35 cycles or until documented progressive disease (PD) occurs. Participants randomized to SOC chemotherapies will be treated with their randomized study drug for up to 4-6 cycles. After this, participants with non-squamous histologies may choose to be treated with maintenance pemetrexed for the remainder of the study or until disease progression, unacceptable adverse event(s) (AEs), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the participant, noncompliance with study treatment or procedures requirements, the participant receives 35 treatments of study treatment (pembrolizumab arm only), or administrative reasons. Participants receiving pembrolizumab who stop drug administration after receiving 35 study treatments for reasons other than disease progression or intolerability, or participants who attain a complete response and stop study treatment may be eligible for retreatment with pembrolizumab upon experiencing disease progression. The decision to retreat with a second course of pembrolizumab will be at the discretion of the Investigator only if participants meet the criteria for retreatment and the study is ongoing. Retreatment (second course) is limited to 17 cycles. Participants randomized to receive SOC chemotherapy may be eligible to receive pembrolizumab if criteria to switch are met.

Switch-Over Phase: This is only applicable for participants randomized to receive SOC. Eligible participants will be treated with pembrolizumab for the remainder of the study or until disease progression, unacceptable AEs, intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the participant, noncompliance with study treatment or procedures requirements, the participant receives 35 treatments of study treatment (pembrolizumab arm only), or administrative reasons.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of Stage IV NSCLC lacking epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) translocation, and received no prior systemic chemotherapy treatment for their metastatic NSCLC
* At least one radiographically measurable lesion per RECIST 1.1
* Life expectancy of at least 3 months
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
* Adequate organ function
* No history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cervical cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy
* Provided newly obtained formalin fixed tumor tissue from a biopsy of a tumor at the time of or AFTER the diagnosis of metastatic disease has been made AND from a site not previously irradiated
* PD-L1 strong expressing tumor as determined by immunohistochemistry (IHC) at a central laboratory
* Female participants must have a negative pregnancy test at screening if of childbearing potential or be of non-childbearing potential
* Female participants of childbearing potential and male partners with female partners of childbearing potential must agree to use 2 adequate barrier methods of contraception during the study and for 120 days after last dose of study drug and up to 180 days after last dose of chemotherapy

Exclusion Criteria:

* EGFR sensitizing mutation and/or ALK translocation
* Has received systemic therapy for the treatment of their stage IV NSCLC. Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of study drug
* Tumor specimen is not evaluable for PD-L1 expression by the central laboratory
* Receiving systemic steroid therapy < 3 days prior to first dose of study drug or receiving any other form of immunosuppressive medication
* Expected to require any other form of systemic or localized antineoplastic therapy during the study
* Received prior systemic cytotoxic chemotherapy, biological therapy, major surgery within 3 weeks of first dose of study drug; received thoracic radiation therapy of > 30 gray (Gy) within 6 months of first dose of study drug
* Received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* Allogenic tissue/solid organ transplant
* Interstitial lung disease or pneumonitis that has required oral or IV steroids
* Received or will receive a live vaccine within 30 days prior to first dose of study drug
* Active infection requiring IV systemic therapy
* Known history of human immunodeficiency virus (HIV)
* Known active tuberculosis, or hepatitis B or C
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Pregnant or breastfeeding, or expecting to conceive or father children during the study and through 120 days after last dose of pembrolizumab or 180 days after last dose of SOC chemotherapy
* Immediate family member who is investigational site or sponsor staff directly involved with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR for the KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1 Positive Non-Small-Cell Lung Cancer . N Engl J Med. 2016;[e published 09 Oct 2016]. doi: 10.1056/NEJMoa1606774
- [Derived] Halmos B, Burke T, Kalyvas C, Insinga R, Vandormael K, Frederickson A, Piperdi B. Indirect comparison of pembrolizumab monotherapy versus nivolumab + ipilimumab in first-line metastatic lung cancer. Immunotherapy. 2022 Apr;14(5):295-307. doi: 10.2217/imt-2021-0273. Epub 2022 Jan 25. PMID 35073727
- [Derived] Satouchi M, Nosaki K, Takahashi T, Nakagawa K, Aoe K, Kurata T, Sekine A, Horiike A, Fukuhara T, Sugawara S, Umemura S, Saka H, Okamoto I, Yamamoto N, Sakai H, Kishi K, Katakami N, Horinouchi H, Hida T, Okamoto H, Atagi S, Ohira T, Rong Han S, Noguchi K, Ebiana V, Hotta K. First-line pembrolizumab vs chemotherapy in metastatic non-small-cell lung cancer: KEYNOTE-024 Japan subset. Cancer Sci. 2021 Dec;112(12):5000-5010. doi: 10.1111/cas.15144. Epub 2021 Nov 5. PMID 34543477
- [Derived] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Derived] Satouchi M, Nosaki K, Takahashi T, Nakagawa K, Aoe K, Kurata T, Sekine A, Horiike A, Fukuhara T, Sugawara S, Umemura S, Saka H, Okamoto I, Yamamoto N, Sakai H, Kishi K, Katakami N, Horinouchi H, Hida T, Okamoto H, Atagi S, Ohira T, Han SR, Noguchi K, Ebiana V, Hotta K. First-line pembrolizumab vs chemotherapy in metastatic non-small-cell lung cancer: KEYNOTE-024 Japan subset. Cancer Sci. 2020 Dec;111(12):4480-4489. doi: 10.1111/cas.14647. Epub 2020 Oct 16. PMID 32926507 (Retraction: PMID 34390097 Cancer Sci. 2021 Aug;112(8):3403)
- [Derived] Lala M, Li TR, de Alwis DP, Sinha V, Mayawala K, Yamamoto N, Siu LL, Chartash E, Aboshady H, Jain L. A six-weekly dosing schedule for pembrolizumab in patients with cancer based on evaluation using modelling and simulation. Eur J Cancer. 2020 May;131:68-75. doi: 10.1016/j.ejca.2020.02.016. Epub 2020 Apr 15. PMID 32305010
- [Derived] Bhadhuri A, Insinga R, Guggisberg P, Panje C, Schwenkglenks M. Cost effectiveness of pembrolizumab vs chemotherapy as first-line treatment for metastatic NSCLC that expresses high levels of PD-L1 in Switzerland. Swiss Med Wkly. 2019 Dec 27;149:w20170. doi: 10.4414/smw.2019.20170. eCollection 2019 Dec 16. PMID 31880807
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Brahmer JR, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Zhang J, Lubiniecki GM, Deitz AC, Rangwala R, Reck M. Health-related quality-of-life results for pembrolizumab versus chemotherapy in advanced, PD-L1-positive NSCLC (KEYNOTE-024): a multicentre, international, randomised, open-label phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1600-1609. doi: 10.1016/S1470-2045(17)30690-3. Epub 2017 Nov 9. PMID 29129441
- [Derived] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, it was planned that participants would be randomized 1:1 to receive either pembrolizumab or investigator-choice standard of care (SOC) chemotherapy and data analysis would be conducted on the two treatment arms: Pembrolizumab and SOC Chemotherapy.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg, administered as intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles or until documented progressive disease (PD) or participant discontinuation.
- SOC Chemotherapy: Participants received 1 of 5 possible standard chemotherapy regimens at the investigator's discretion by IV infusion: paclitaxel 200 mg/m^2 and carboplatin Area Under the Curve (AUC) 5 or 6, administered on Day 1 of each 21-day cycle for 4-6 cycles; pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6, on Day 1 of each 21-day cycle for 4-6 cycles; pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, on Day 1 of each 21-day cycle for 4-6 cycles; gemcitabine 1250 mg/m^2, administered on Days 1 and 8 of each 21-day cycle and carboplatin AUC 5 or 6, on Day 1 of a 21-day cycle, for 4-6 cycles; gemcitabine 1250 mg/m^2, on Days 1 and 8 of each 21-day cycle and cisplatin 75 mg/m^2, on Day 1 of each 21-day cycle for 4-6 cycles or until documented PD or participant discontinuation. Participants with documented disease progression following chemotherapy can switch to receive pembrolizumab for up to 35 cycles (approximately 2 years). Eligible participants who switched to and then stopped pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 additional year).
Period: Overall Study
Arm/Group | Pembrolizumab | SOC Chemotherapy
Started | 154 | 151
Treated | 154 | 150
Chemotherapy Switch to Pembrolizumab | 0 | 83
Second Course Pembrolizumab | 12 | 1
Completed | 0 | 0
Not Completed | 154 | 151
Not completed — Adverse Event | 13 | 9
Not completed — Death | 92 | 112
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Follow up ended by sponsor | 43 | 20

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg, administered as IV infusion on Day 1 of each 21-day cycle for up to 35 cycles or until documented PD or participant discontinuation.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | SOC Chemotherapy | Total
Number analyzed (Participants) | 154 | 151 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (10.1) | 64.6 (9.5) | 64.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 56 | 118
  Male | 92 | 95 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 148 | 135 | 283
  Unknown or Not Reported | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 25 | 21 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 125 | 126 | 251
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) Status (0, 1 or 2) [Number; unit: Rating] — Eastern Cooperative Oncology Group (ECOG) Performance. ECOG is presented where 0 = Fully active, no performance restrictions; 1 = Strenuous physical activity restricted, fully ambulatory & able to carry out light work; and 2 = In bed <50% of the time, ambulatory and capable of all self-care, but unable to carry out any work activities.
  Rating
    ECOG = 0 | 54 | 53 | 107
    ECOG = 1 | 99 | 98 | 197
    ECOG = 2 | 1 | 0 | 1
Histology [Number; unit: Participants] — Participants were categorized according to the histology of their carcinoma
  Participants
    ADENOCARCINOMA | 104 | 108 | 212
    ADENOSQUAMOUS | 2 | 2 | 4
    LARGE CELL CARCINOMA | 2 | 2 | 4
    NON-SQUAMOUS CELL CARCINOMA | 5 | 7 | 12
    POORLY DIFFERENTIATED | 9 | 3 | 12
    SARCOMATOID | 3 | 2 | 5
    SQUAMOUS CELL CARCINOMA | 29 | 26 | 55
    POORLY DIFFERENTIATED SQUAMOUS CELL CARCINOMA | 0 | 1 | 1
Geographic Region of Enrolling Site [Count of Participants; unit: Participants] — Count of Participants enrolled in sites in Non-East Asia and East Asia
  Participants
    Non-East Asia | 133 | 132 | 265
    East Asia | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at Month 6
Description: PFS was defined as the time from randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on blinded independent central radiologists' (BICR) review. Progressive Disease (PD) was defined as ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. (Note: the appearance of one or more new lesions was also considered progression). Participants were evaluated every 9 weeks with radiographic imaging to assess their response to treatment. The data cutoff was 09-May-2016. The PFS rate at Month 6 was calculated.
Time Frame: Month 6
Population: The Intention-to-treat (ITT) population included all randomized participants. Participants were included in the treatment group to which they were randomized, regardless of whether or not they received study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | SOC Chemotherapy
Number analyzed (Participants) | 154 | 151
Percentage of Participants | 62.1 [53.8 to 69.4] | 50.3 [41.9 to 58.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs SOC Chemotherapy; Test type: Superiority or Other; p < 0.001, Regression, Cox — One-sided p-value based on log-rank test; Treatment as a covariate stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1) and histology (squamous vs. nonsquamous); Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.37 to 0.68]

2. Secondary Outcome: Overall Survival (OS) Rate
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The data cutoff was 10-July-2017. The median OS rate at 12 months is presented.
Time Frame: 12 months
Population: The ITT population included all randomized participants. Participants were included in the treatment group to which they were randomized, regardless of whether or not they received study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | SOC Chemotherapy
Number analyzed (Participants) | 154 | 151
Percentage of Participants | 70.3 [62.3 to 76.9] | 54.8 [46.4 to 62.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs SOC Chemotherapy; Test type: Superiority or Other; p = 0.002, Regression, Cox — One-sided p-value based on log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.47 to 0.86]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. ORR was assessed from enrollment/treatment initiation of a participant through data cutoff of 09-May-2016. The ORR is presented for each treatment group.
Time Frame: Up to ~1.6 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | SOC Chemotherapy
Number analyzed (Participants) | 154 | 151
Percentage of Participants | 44.8 [36.8 to 53.0] | 27.8 [20.8 to 35.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs SOC Chemotherapy; H0: difference in %=0 vs. H1: difference in % >0; Test type: Superiority or Other; p = 0.0011, Miettinen & Nurminem method — One-sided p-value for testing; Stratified by geographic region (East Asia vs. non-East Asia), ECOG PS (0 vs. 1) and histology (squamous vs. nonsquamous); Difference in percentages = 16.6, 95% CI 2-sided [6.0 to 27.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 80 months.
Description: All-cause mortality: All randomized participants. Safety: All randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression" and "Malignant neoplasm progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg, administered as intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles or until documented progressive disease (PD) or participant discontinuation.
- SOC Chemotherapy First Course: Participants received 1 of 5 possible standard chemotherapy regimens at the investigator's discretion by IV infusion: paclitaxel 200 mg/m^2 and carboplatin Area Under the Curve (AUC) 5 or 6, administered on Day 1 of each 21-day cycle for 4-6 cycles; pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6, on Day 1 of each 21-day cycle for 4-6 cycles; pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2, on Day 1 of each 21-day cycle for 4-6 cycles; gemcitabine 1250 mg/m^2, administered on Days 1 and 8 of each 21-day cycle and carboplatin AUC 5 or 6, on Day 1 of a 21-day cycle, for 4-6 cycles; gemcitabine 1250 mg/m^2, on Days 1 and 8 of each 21-day cycle and cisplatin 75 mg/m^2, on Day 1 of each 21-day cycle for 4-6 cycles or until documented PD or participant discontinuation. Participants with documented disease progression following chemotherapy can switch to receive pembrolizumab for up to 35 cycles (approximately 2 years). Eligible participants who switched to and then stopped pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 additional year).
- SOC Chemotherapy Switched Over to Pembrolizumab First Course: Qualified participants who received the SOC chemotherapy first course but continued to experience disease progression, at the investigator's discretion, initiated a course of pembrolizumab IV 200 mg, every cycle (three weeks) for up to 35 cycles up to ~2 years.
- Pembrolizumab Second Course: Qualified participants who received the pembrolizumab first course and achieved CR, PR, or stable disease, and progressed after discontinuation, at the investigator's discretion, initiated a second course of pembrolizumab at the same dose and schedule for up to 17 cycles (approximately 1 additional year).
- SOC Switched Over to Pembrolizumab Second Course: One qualified participant received SOC chemotherapy first course, but continued to experience disease progression and at investigator's discretion switched to a course of pembrolizumab IV 200 mg, every cycle (three weeks) for up to 35 cycles up to ~2 years. The participant then initiated a second course of pembrolizumab at the same dose and schedule for up to ~1 additional year until documented PD or participant discontinuation.
Arm/Group | Pembrolizumab First Course | SOC Chemotherapy First Course | SOC Chemotherapy Switched Over to Pembrolizumab First Course | Pembrolizumab Second Course | SOC Switched Over to Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 103/154 | 60/151 | 62/83 | 4/12 | 1/1
Serious Adverse Events (participants affected / at risk) | 79/154 | 70/150 | 27/83 | 2/12 | 0/1
Other Adverse Events (participants affected / at risk) | 140/154 | 142/150 | 72/83 | 10/12 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=154) | SOC Chemotherapy First Course (N=150) | SOC Chemotherapy Switched Over to Pembrolizumab First Course (N=83) | Pembrolizumab Second Course (N=12) | SOC Switched Over to Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 13 (13) | 2 (2) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood corticotrophin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brown-Sequard syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertensive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=154) | SOC Chemotherapy First Course (N=150) | SOC Chemotherapy Switched Over to Pembrolizumab First Course (N=83) | Pembrolizumab Second Course (N=12) | SOC Switched Over to Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 24 (28) | 77 (98) | 4 (4) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 10 (17) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 35 (67) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 18 (32) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 10 (11) | 2 (3) | 5 (7) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 16 (16) | 3 (3) | 8 (8) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 14 (17) | 10 (10) | 7 (7) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 7 (13) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 35 (43) | 33 (54) | 7 (7) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 41 (65) | 33 (43) | 18 (22) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 9 (14) | 3 (3) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 33 (44) | 68 (129) | 15 (19) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 8 (8) | 17 (23) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (20) | 36 (65) | 8 (9) | 0 (0) | 0 (0)
Asthenia (General disorders) | 12 (17) | 17 (30) | 7 (7) | 0 (0) | 0 (0)
Chest pain (General disorders) | 16 (17) | 16 (16) | 5 (6) | 0 (0) | 0 (0)
Fatigue (General disorders) | 37 (45) | 53 (93) | 18 (19) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (7) | 3 (4) | 1 (1) | 0 (0)
Malaise (General disorders) | 6 (6) | 12 (13) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 19 (20) | 15 (19) | 3 (4) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 27 (36) | 14 (16) | 8 (8) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 8 (9) | 4 (5) | 5 (6) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (27) | 2 (2) | 9 (10) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (18) | 5 (7) | 9 (12) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (11) | 8 (11) | 4 (4) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 4 (4) | 3 (5) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (20) | 11 (15) | 4 (4) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 15 (19) | 7 (9) | 4 (4) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 10 (14) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 12 (15) | 21 (26) | 5 (9) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 21 (37) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 19 (28) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 14 (15) | 11 (12) | 6 (8) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 17 (25) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 33 (36) | 49 (71) | 12 (13) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (17) | 9 (10) | 2 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (9) | 6 (7) | 3 (4) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (8) | 7 (7) | 3 (6) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7) | 13 (18) | 5 (5) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (17) | 12 (13) | 7 (8) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (47) | 17 (21) | 16 (18) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (26) | 18 (21) | 4 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (12) | 10 (13) | 6 (8) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 20 (25) | 12 (16) | 5 (7) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 13 (13) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (17) | 7 (8) | 7 (7) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 10 (10) | 3 (3) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 16 (18) | 11 (11) | 7 (7) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (44) | 21 (24) | 16 (17) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (50) | 24 (29) | 9 (10) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 5 (5) | 7 (10) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (12) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 15 (15) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (18) | 1 (1) | 7 (7) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (46) | 6 (6) | 13 (13) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 28 (43) | 7 (8) | 8 (13) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (2) | 6 (6) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 11 (13) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 4 (4) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02142738/Prot_SAP_000.pdf